CLINICAL TRIAL: NCT04638816
Title: A Study Comparing Hyaluronic Acid Effectiveness & Evaluating Cheek Results With Restylane
Brief Title: Study to Evaluate Satisfaction After Treatment With Restylane
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05DF2004
Record Dates: First submitted 2020-11-16; First posted 2020-11-20 (Actual); Results first posted 2024-03-06 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2023-08

CONDITIONS: Cheek Augmentation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Restylane Volyme (Experimental): Hyaluronic Acid
  Interventions: Device: Restylane Volyme
- Restylane Lyft Lidocaine (Experimental): Hyaluronic Acid
  Interventions: Device: Restylane Lyft Lidocaine

INTERVENTIONS:
Device: Restylane Volyme — Hyaluronic Acid: Injectable gel for contouring effect (of cheek volumization).
  Arms: Restylane Volyme
Device: Restylane Lyft Lidocaine — Hyaluronic Acid: Injectable gel for projection effect (of cheek augmentation).
  Arms: Restylane Lyft Lidocaine

SUMMARY:
Open-label, phase IV, post-marketing study to evaluate aesthetic improvement and satisfaction after treatment with Restylane

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent to participate in the study
* Adult women who intend to undergo cheek augmentation

Exclusion Criteria:

* Subjects presenting with known allergy to HA (hyaluronic acid) filler or amide local anesthetics
* Subjects with a previous implant other than HA in or near the intended treatment site
* Participation in any other clinical study within three (3) months before treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female adult subject.
Enrollment: 60 (Actual)
Dates: Start 2021-04-16 (Actual); Primary Completion 2021-07-03 (Actual); Study Completion 2021-08-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Galderma R&D
Locations (3):
- Canada (3):
  - Galderma Study Site, Vancouver, British Columbia
  - Galderma Study Site, Woodbridge, Ontario
  - Galderma Study Site, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Restylane Volyme | Restylane Lyft Lidocaine
Started | 30 | 30
Completed | 30 | 28
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Restylane Volyme | Restylane Lyft Lidocaine | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Full Range); unit: years] | 48.8 [24 to 77] | 49 [23 to 69] | 48.9 [23 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 30 | 60
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 29 | 29 | 58
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 26 | 29 | 55
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  Canada | 30 | 30 | 60
Fitzpatrick Skin Type (FST) [Count of Participants; unit: Participants] — I (white, very fair, red or blond hair, blue eyes, freckles), II (white, fair, red or blond hair; blue, hazel or green eyes), III (cream white, fair with any eye or hair color, very common), IV (brown, typical Mediterranean Caucasian skin), V (dark brown, Middle Eastern skin type), VI (black)
  Participants
    FST I | 1 | 0 | 1
    FST II | 10 | 7 | 17
    FST III | 12 | 15 | 27
    FST IV | 7 | 7 | 14
    FST V | 0 | 1 | 1
    FST VI | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Assess Treatment With Restylane Volyme and Restylane Lyft Lidocaine Using GAIS
Description: The 7-grade Global Aesthetic Improvement Scale (GAIS) assess the appearance of the treatment area (cheeks) compared to pre-treatment. The rating is very much improved, much improved, improved, no change, worse, much worse, or very much worse.
Time Frame: 4 weeks after last treatment, up to 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Restylane Volyme | Restylane Lyft Lidocaine
Number analyzed (Participants) | 30 | 29
Participants
  Very much improved | 20 | 17
  Much improved | 9 | 9
  Improved | 1 | 3
  No change | 0 | 0
  Worse | 0 | 0
  Much worse | 0 | 0
  Very much worse | 0 | 0

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | Restylane Volyme | Restylane Lyft Lidocaine
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 1/30 | 1/30
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Restylane Volyme (N=30) | Restylane Lyft Lidocaine (N=30)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PIs agree not to present or publish any data or reports collected individually or by subgroup of sites prior to full, initial publication based on all data obtained from all sites.

DOCUMENTS (2):
  • Study Protocol (2020-11-03): https://cdn.clinicaltrials.gov/large-docs/16/NCT04638816/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-23): https://cdn.clinicaltrials.gov/large-docs/16/NCT04638816/SAP_001.pdf